CLINICAL TRIAL: NCT01318915
Title: Immunosuppression With Antithymocyte Globulin, Rituximab, Tacrolimus, Mycophenolate Mofetil and Sirolimus, Followed by Withdrawal of Immunosuppression, in Living-donor Renal Transplant Recipients
Brief Title: Research Study of ATG and Rituximab in Renal Transplantation
Acronym: RESTARRT
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The stopping rule for incidence of acute rejection was met.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN039ST
Record Dates: First submitted 2011-03-15; First posted 2011-03-21 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Renal Transplant Recipients
Keywords: Kidney transplantation; Living donor transplant; Graft rejection; Graft loss; Induction with rituximab and ATG; Immunosuppression (IS)
MeSH Terms: interventions — thymoglobulin; Antilymphocyte Serum; Rituximab; Tacrolimus; Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Induction (Rituximab and ATG) (Experimental): Study participants will undergo induction with rituximab and ATG and an initial maintenance therapy with tacrolimus, mycophenolate mofetil (MMF) and sirolimus. MMF will be discontinued on day 12. Participants will be evaluated for eligibility for tacrolimus withdrawal which must be initiated between weeks 26 and 38. Tacrolimus withdrawal must be completed in no fewer than 4 weeks and no more than 8 weeks. Then after at least 26 weeks on sirolimus monotherapy, participants will be evaluated for eligibility for sirolimus withdrawal which must be initiated between weeks 56 and 88. Sirolimus withdrawal must be completed in no fewer than 12 weeks and no more than 26 weeks.
  Interventions: Drug: ATG; Drug: Rituximab; Drug: Tacrolimus; Drug: Sirolimus; Drug: MMF

INTERVENTIONS:
Drug: ATG — 1.5 mg/kg IV infusion on day of transplant, and 3 additional on days 2 through 7 after transplant.
  Other Names: Thymoglobulin; Antithymocyte globulin
Drug: Rituximab — 375 mg/m^2 IV infusion on day -6 before transplant and on day 1 after transplant.
  Other Names: Rituxan
Drug: Tacrolimus — Taken orally. Tacrolimus dose adjusted to maintain target blood levels of 6-10 ng/mL.
  Other Names: Prograf; FK-506; Fujimycin
Drug: Sirolimus — Taken orally. Initial dose, 2 mg daily on day 10 post-transplant, subsequently adjusted to achieve trough levels of 8-12 ng/mL through week 56. Sirolimus withdrawal will be initiated between week 56 and week 88 in eligible participants.
  Other Names: Rapamune; Rapamycin
Drug: MMF — 1 g twice daily on days 0 through 12
  Other Names: mycophenolate mofetil

SUMMARY:
The purpose of this study is see if a combination of two drugs, (ATG and rituximab), given at the time of the transplant surgery, will help reduce or eliminate the need for long term immunosuppressive medication.

DETAILED DESCRIPTION:
Kidneys remove excess fluid and waste from the blood. When kidneys lose their filtering ability, dangerous levels of fluid and waste accumulate in the body - a condition known as kidney failure. There are two ways to treat kidney failure. One way is to get dialysis indefinitely. The second way is to get a kidney transplant. A kidney transplant is often the best treatment for kidney failure. A kidney transplant is a surgical procedure to place a healthy kidney from a donor into a person whose kidneys no longer function properly. This study is for people who will receive a kidney transplant from a very well matched, living blood relative. The immune system is the body's defense system against illness. After transplant, the immune system will think that the new kidney is a foreign invader and will try to attack or reject the transplanted kidney. Immunosuppressive drugs protect the transplanted kidney by suppressing the immune system. People who have kidney transplants must take immunosuppressive drug for the rest of their lives. If they stop, their immune system may reject the transplanted kidney. Immunosuppressive drugs make it hard for the body to fight off infections. In addition, they can cause high blood pressure, kidney damage, plaque build-up in the blood vessels, high cholesterol, diabetes and bone disease. They may also make the body more likely to get some types of cancer (mainly cancer of the white blood cells and/or skin) and other serious side effects.

Because of the side effects of immunosuppressive drugs, an important goal of transplant research is to allow people to accept their transplanted organ without always having to take immunosuppressive drugs. This is called tolerance. The RESTARRT study is testing a combination of two medications, rituximab and anti-thymocyte globulin (ATG), to see if they can help people reduce or eliminate the need for life-long immunosuppressive medications. ATG has been used for over 10 years to treat transplant rejection; rituximab is used to treat rheumatoid arthritis and two types of cancer. ATG works on immune cells called 'T cells' that are involved in transplant rejection, while rituximab works on a different type of cell called 'B cells.' Researchers hope that targeting both these cell types at the same time will help reset the immune system so that it accepts the transplanted kidney.

Frequent visits are required during the first two months of the study. Then, study visits take place about every 4 weeks, but more often (every 2 weeks) when reducing medication doses. After two years, participants will be asked to return for check-ups every 3 months. Study visits may include consultations with the transplant doctors, physical exam, blood and/or urine samples and kidney biopsies at several times during the study. In all, participation could last up to 4 years. All study-related medications and tests are provided at no charge to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a first renal allograft from a single haplotype matched or greater living related donor who is no older than 65, or a second degree relative with an Human Leukocyte Antigen(HLA) type that is consistent with a single haplotype match with the recipient.
* Demonstration of absence of anti-HLA antibodies using solid phase micro particle technology (by Luminex® phenotype panel or Luminex single antigen bead test) performed 7 days or less prior to the first dose of rituximab, as assessed by local laboratories.No evidence of anti-HLA antibodies in current or past sera.Negative T- and B-cell crossmatch as determined by flow cytometric assay measured 7 days or less prior to the first dose of rituximab.
* Single-organ recipients (kidney only).
* Serologic evidence of prior exposure to Epstein-Barr virus (EBV).
* For women of childbearing potential: a negative serum or urine pregnancy test with sensitivity less than 50 mIU/m within 72 hours before the start of study medication.
* Use of FDA-approved methods of contraception (those with less than a 5% failure rate) by all participants from the time that study treatment begins until 104 weeks (24 months) after renal transplantation.
* Ability to receive oral medication.
* Ability to understand and provide informed consent.

Exclusion Criteria:

* Recipient of a kidney from a donor who is older than 65 years.
* History of cancer within the last 5 years, except for nonmelanoma skin cell cancers cured by local resection and cervical carcinoma in situ.
* Women who are breastfeeding.
* Uncontrolled hyperlipidemia (total serum cholesterol more than 300 mg/dL and/or triglycerides more than 400 mg/dL).
* Platelet count less than 100,000/μL at study entry.
* Seropositivity for HIV-1, Hepatitis C virus (HCV) (confirmed by HCV PCR), hepatitis B surface antigen, or Hepatitis B virus (HBV) core antibody (confirmed by HBV PCR).
* Active tuberculosis (TB) within the previous 3 years regardless of treatment history for TB. Participants with a known positive purified protein derivative (PPD) or positive Quantiferon assay will not be eligible for the study unless they have completed treatment for latent TB and have a negative chest x-ray at the time of enrollment. PPD testing or Quantiferon testing done within 52 weeks before transplant is acceptable as long as there is documentation of the results. Prior recipients of a Bacille Calmette-Guérin vaccination (BCG) are not exempt.
* Underlying renal disease with a high risk of disease recurrence in the transplanted kidney, including focal segmental glomerulosclerosis, types I or II membranoproliferative glomerulonephritis, and hemolytic-uremic syndrome/thrombotic thrombocytopenic purpura.
* The presence of any medical condition that the investigator deems incompatible with participation in the trial.
* Known sensitivity to antithymocyte globulin, rituximab, tacrolimus, sirolimus, MMF, or corticosteroids.
* Current use of systemic corticosteroids or antibody-based therapies (e.g., infliximab, adalimumab, or etanercept).
* Use of any investigational drug within 30 days of transplantation.
* Receipt of a live vaccine within 3 months of enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07-25; Primary Completion 2016-06-17 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Markmann, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rogosin Institute/New York Presbyterian-Cornell, New York, New York
  - Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The plan is to provide data access to the public in the Immunology Database and Analysis Portal (ImmPort, http://www.immport.org/). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: After completion of the study.
Access Criteria: Will be available to the public.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- [Background] Solez K, Colvin RB, Racusen LC, Haas M, Sis B, Mengel M, Halloran PF, Baldwin W, Banfi G, Collins AB, Cosio F, David DS, Drachenberg C, Einecke G, Fogo AB, Gibson IW, Glotz D, Iskandar SS, Kraus E, Lerut E, Mannon RB, Mihatsch M, Nankivell BJ, Nickeleit V, Papadimitriou JC, Randhawa P, Regele H, Renaudin K, Roberts I, Seron D, Smith RN, Valente M. Banff 07 classification of renal allograft pathology: updates and future directions. Am J Transplant. 2008 Apr;8(4):753-60. doi: 10.1111/j.1600-6143.2008.02159.x. Epub 2008 Feb 19. PMID 18294345
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction (Rituximab and ATG): Adult living donor kidney transplant recipients were enrolled into the study prior to transplant. Participants received a novel induction regimen of ATG and rituximab that included 4 doses of ATG 1.5 mg/kg and 2 doses of rituximab 375 mg/m^2. The first dose of rituximab was given ~ day -6 pre-transplant, and the second dose on day 1-3 post-transplant. The first dose of ATG was given on the day of transplant, with the additional three doses administered on days 2-7 post-transplant (not on the same day as rituximab). Participants were maintained on anti-rejection medications tacrolimus, MMF, and sirolimus post-transplant. Participants were evaluated for eligibility to proceed with immunosuppressive maintenance withdrawal (IMW), a gradual withdrawal of their anti-rejection medications, starting as early as 26 weeks post-transplant. IMW for eligible participants proceeded with close monitoring per protocol over a period of 68-104 weeks.
Period: Overall Study
Arm/Group | Induction (Rituximab and ATG)
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] — Serum creatinine provides an estimate of how well the kidneys filter (glomerular filtration rate). Higher results= poorer kidney function. The baseline creatinine interval per protocol is defined as the 2 to 4 week interval post-kidney transplant and is calculated using the lowest N=3 serum creatinine values during this pre-defined interval, the interval prior to immunosuppressive maintenance withdrawal (IMW) initiation. Normal values: Adult males, 0.7 to 1.3 mg/dL; adult females, 0.6 to 1.1 mg/dL.
  mg/dL | 1.7 (0.73)
eGFR [Mean (Standard Deviation); unit: mg/dL] — Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. The equation developed by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) is used to estimate GFR (e.g., eGFR) from serum creatinine. Baseline serum creatinine was used in the equation, which is the average of the lowest three creatinine values during 2 to 4 weeks post-transplant, excluding days on dialysis.
  mg/dL | 55.1 (20.79)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — The systolic blood pressure collected on the day of transplant. If there is no value recorded on the day of transplant, the value from the screening visit is used. Systolic blood pressure measures the pressure on the blood vessels when the heart is beats and thus is pushing blood to the rest of the body. A normal systolic blood pressure is lower than 120 mmHg. High blood pressure, also known as hypertension, is a risk factor for coronary artery disease, stroke, heart failure, and other complications if left unmanaged.
  mmHg | 142.3 (21.27)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — The diastolic blood pressure collected on the day of transplant. If there is no value recorded on the day of transplant, the value from the screening visit is used. Diastolic blood pressure measures the pressure in the arteries when the heart is at rest and is thus filled with blood. A normal diastolic blood pressure is lower than 80 mmHg. High blood pressure, as known as hypertension, is a risk factor for coronary artery disease, stroke, heart failure, and other complications if left unmanaged.
  mmHg | 82.5 (15.01)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — The total cholesterol collected on the day of transplant. If there is no value recorded on the day of transplant, the value from the screening visit is used. Total cholesterol measures the amount of cholesterol found in the blood. Cholesterol is a waxy substance your body needs to build cells, but too much can be a problem since it can build-up in arteries. Narrowed arteries can result in heart attack or stroke. A value less than 200 mg/dL is considered good.
  mg/dL | 181.6 (67.10)
Glucose [Mean (Standard Deviation); unit: mg/dL] — The glucose collected on the day of transplant. If there is no value recorded on the day of transplant, the value from the screening visit is used. Glucose, a sugar, is an energy source that the body relies on to properly function. If levels are too high for a long period of time, diabetes can develop. Diabetes can result in many long-term complications such as eye, kidney, and nerve damage, stroke, and cardiovascular complications. Fasting levels for glucose should be around 70-99 mg/dL and less than 140 mg/dL within 2 hours after a meal.
  mg/dL | 102.0 (22.57)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Successfully Withdrawn From Immunosuppression and Remained Off Immunosuppression for at Least 52 Weeks
Description: Participants are considered successfully withdrawn from immunosuppression if they remained off immunosuppression for at least 52 weeks without evidence of rejection, as determined by a biopsy performed 52 weeks after completion of immunosuppression withdrawal. All participants who failed to complete immunosuppression withdrawal, regardless of reason, or failed to have a biopsy 52 weeks after completion of immunosuppression withdrawal, were considered to have failed. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through 52 weeks after discontinuation of all immunosuppression
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 20 [2.5 to 55.6]

2. Secondary Outcome: Percent of Transplanted Participants Who Remain Off Immunosuppression for at Least 52 Weeks Including Those in Whom the 52 Week Biopsy Was Not Performed
Description: Participants are considered successfully withdrawn from immunosuppression if they remained off immunosuppression for at least 52 weeks without evidence of rejection. A biopsy performed 52 weeks after completion of immunosuppression withdrawal confirmed that there was no sub-clinical evidence of rejection. This result considers a participant off all immunosuppression for at least 52 weeks with or without the confirmatory week 52 biopsy as a success. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through 52 weeks after discontinuation of all immunosuppression
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 20 [2.5 to 55.6]

3. Secondary Outcome: Percent of Transplanted Participants Who Remain Off Immunosuppression for the Duration of the Study as Defined as Completion of All Schedules of Events/Followed Through August 25, 2017
Description: Participants that remained off all immunosuppression through the completion of study participation. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through study completion (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 10 [0.3 to 44.5]

4. Secondary Outcome: Percent of Transplanted Participants Who Achieve Sirolimus Monotherapy Within 52 Weeks Post-transplant
Description: Participants that were treated with only sirolimus within 52 weeks after transplantation in those who could tolerant sirolimus. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through 52 weeks post-transplantation
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study that tolerated sirolimus
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 7
Percent of participants | 86 [42.1 to 99.6]

5. Secondary Outcome: Percent of Transplanted Participants Who Achieve MMF or Mycophenolic Acid Monotherapy Within 52 Weeks Post-transplant in Those Participants Intolerant of Sirolimus
Description: Participants that were treated with only mycophenolate mofetil (MMF) or mycophenolic acid within 52 weeks after transplantation in those who could not tolerate sirolimus. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through 52 weeks post-transplantation
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study that could not tolerate sirolimus
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 3
Percent of participants | 33 [0.8 to 90.6]

6. Secondary Outcome: Percent of Transplanted Participants Who Achieve Either Sirolimus Monotherapy or Monotherapy on a Mycophenolic Compound Within 52 Weeks Post-transplant
Description: Participants that were treated with only sirolimus or treated with only mycophenolate mofetil (MMF) or mycophenolic acid within 52 weeks after transplantation. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through 52 weeks post-transplantation
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 70 [34.8 to 93.3]

7. Secondary Outcome: Immunosuppression-free Duration in Days, Defined as Time From Completion of Immunosuppression Withdrawal to End of Trial Participation or to Time of Restarting Immunosuppression
Description: Time (in days) from when the participant is off all immunosuppression to the end of trial participation or re-initiation of immunosuppression, whichever is earliest.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study that stopped using all immunosuppression drugs
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Transplanted: Adult living donor kidney transplant recipients that were enrolled into the study prior to transplant and met all criteria for study participation. These participants received a novel induction regimen of ATG and rituximab that included 4 doses of ATG 1.5 mg/kg and 2 doses of rituximab 375 mg/m^2. The first dose of rituximab was given ~day -6 prior to transplant, and the second dose was given on day 1-3 post-transplant. The first dose of ATG was given on the day of transplant, with the additional three doses administered on days 2-7 post-transplant (not on the same day as rituximab). Participants were maintained on the anti-rejection medications tacrolimus, MMF, and sirolimus after transplant. Participants were evaluated for eligibility to start gradual withdrawal of their anti-rejection medications starting as early as 26 weeks post-transplant. Eligible participants were gradually withdrawn from anti-rejection medication over a period of 68-104 weeks.
Arm/Group | Transplanted
Number analyzed (Participants) | 6
Days | 374 [198 to 639]

8. Secondary Outcome: Time From Completion of Immunosuppression Withdrawal to First Episode of Acute Rejection or Presumed Acute Rejection
Description: Time (in days) from when the participant is off all immunosuppression to the first episode of biopsy proven or presumed acute rejection.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study that stopped using all immunosuppression drugs and had acute rejection or presumed acute rejection.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Induction (Rituximab and ATG): Adult living donor kidney transplant recipients were enrolled into the study prior to transplant. Participants received a novel induction regimen of ATG and rituximab that included 4 doses of ATG 1.5 mg/kg and 2 doses of rituximab 375 mg/m^2. The first dose of rituximab was given ~day -6 pre-transplant, and the second dose was given on day 1-3 post-transplant. The first dose of ATG was given on the day of transplant, with the additional three doses administered on days 2-7 post-transplant (not on the same day as rituximab). Participants were maintained on anti-rejection medications tacrolimus, MMF, and sirolimus post-transplant. Participants were evaluated for eligibility to proceed with immunosuppressive maintenance withdrawal (IMW), a gradual withdrawal of their anti-rejection medications, starting as early as 26 weeks post-transplant. IMW for eligible participants proceeded with close monitoring per protocol over a period of 68-104 weeks.
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 5
Days | 380 [198 to 452]

9. Secondary Outcome: Time From Completion of Immunosuppression Withdrawal to First Diagnosis of Chronic T Cell Mediated or Antibody-mediated Rejection
Description: Time (in days) from the time the participant is off all immunosuppression to the first episode of chronic T cell mediated or chronic antibody-mediated rejection. This assessment also includes progressive interstitial fibrosis/tubular atrophy (IF/TA), transplant glomerulopathy or chronic obliterative arteriopathy without an alternative, non-rejection related cause.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study that stopped using all immunosuppression drugs and were diagnosed with chronic rejection.
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 0

10. Secondary Outcome: Percent of Transplanted Participants With Graft Loss
Description: A participant is considered to have graft loss when the donated kidney needs to be removed, the participant is retransplanted with another donor kidney, or chronic dialysis is instituted. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 0 [0 to 30.9]

11. Secondary Outcome: Percent of Transplant Participants Who Died
Description: Death after receiving a kidney transplant. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 0 [0 to 30.9]

12. Secondary Outcome: Percent of Transplanted Participants With Acute Rejection or Presumed Acute Rejection
Description: Participants with either biopsy proven acute rejection per Banff guidelines or participants that were treated for acute rejection in the absence of a biopsy. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 90 [55.5 to 99.8]

13. Secondary Outcome: Histological Severity of Biopsies Demonstrating Acute Rejection as Measured by Banff 2007 Grade
Description: Biopsy-confirmed 1.) acute cellular rejection and 2.) acute antibody-mediated rejection was classified according to Banff 2007 criteria of renal allograft pathology for renal allograft rejection. A Banff result of indeterminate was not classified as rejection.
  Acute cellular rejection occurs when lesions at the site of the graft characteristically are infiltrated with large numbers of lymphocytes and macrophages that cause tissue damage. Acute cellular rejection is defined as a grade ≥ IA. Severity is graded as IA, IB, IIA, IIB, or III, with IA being the mildest form of cellular rejection and III being the most severe.
  Acute antibody-mediated rejection-or humoral rejection-is defined as a grade ≥1. Severity is graded as I, II, or III, with I being the mildest form of antibody-mediated rejection and III being the most severe.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study.
Measure: Number; unit: Biopsies
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Biopsies
  Acute Cellular Rejection (Type IA) | 7
  Acute Cellular Rejection (Type IB) | 3
  Acute Cellular Rejection (Type IIA) | 0
  Acute Cellular Rejection (Type IIB) | 0
  Acute Cellular Rejection (Type III) | 0
  Acute Antibody-Mediated Rejection (Type I) | 0
  Acute Antibody-Mediated Rejection (Type II) | 0
  Acute Antibody-Mediated Rejection (Type III) | 0

14. Secondary Outcome: Percent of Participants With Chronic T Cell-mediated or Antibody-mediated Rejection
Description: This assessment included participants who experienced chronic T cell-mediated rejection or chronic antibody mediated rejection as well as progressive interstitial fibrosis/tubular atrophy (IF/TA), transplant glomerulopathy or chronic obliterative arteriopathy without an alternative, non-rejection-related cause.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 0 [0 to 30.9]

15. Secondary Outcome: Time From Transplant to the First Episode of Acute Rejection Requiring Treatment
Description: Time (in days) from transplant to the start date of the first dose of treatment for acute rejection. This includes acute rejection episodes requiring treatment that are not biopsy proven.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study that had acute rejection requiring treatment.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 6
Days | 1008.5 [577 to 1139]

16. Secondary Outcome: Percent of Participants Requiring Anti-lymphocyte Therapy (OKT3, ATG) for an Acute Rejection Event
Description: Anti-lymphocyte therapy is a drug that targets specific cells in the immune system called lymphocytes (white blood cells). This therapy helps stop the participant's immune system from attacking the donor kidney. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Percent of participants | 20 [2.5 to 55.6]

17. Secondary Outcome: Number of Adverse Events, Including Number of Post-transplant Infections, Wound Complications, Lymphocoele, Post-transplant Diabetes Mellitus, and Malignancies
Description: Adverse events that are reported as being a post-transplant infection, wound complication, lymphocoele (a collection of fluid in the lymphatic system), post-transplant diabetes mellitus or malignancy.
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant)
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study
Measure: Number; unit: Events
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
Events
  Post-Transplant Infection | 4
  Wound Complications | 1
  Lymphocoele | 0
  Post-Transplant Diabetes Mellitus | 0
  Malignancy | 0

18. Secondary Outcome: Participant Renal Function as Measured by GFR Using CKD-EPI
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. A value less than 15 indicates kidney failure, 15 to 29 indicates severe loss of kidney function, 30 to 44 indicates moderate to severe loss of kidney function, 45 to 59 mild to moderate loss of kidney function, 60 to 89 indicates mild loss of kidney function, and 90 or higher indicates normal kidney function. The equation developed by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) is used to estimate GFR from serum creatinine. The value closest to and within 6 weeks of the day expected was selected.
Time Frame: 26, 52, 104, 156, and 208 Weeks Post-Transplant
Population: Participants that received induction (Rituximab and ATG) and were transplanted on study, with data available at each time point.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m^2
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
mL/min/1.73m^2
  26 Weeks Post-Transplant | 60.3 [57.1 to 64.3]
  52 Weeks Post-Transplant | 70.9 [57.0 to 74.6]
  104 Weeks Post-Transplant: number analyzed (Participants) | 7
  104 Weeks Post-Transplant | 63.7 [58.6 to 69.5]
  156 Weeks Post-Transplant: number analyzed (Participants) | 4
  156 Weeks Post-Transplant | 56.7 [54.9 to 85.6]
  208 Weeks Post-Transplant: number analyzed (Participants) | 4
  208 Weeks Post-Transplant | 56.0 [37.5 to 94.1]

19. Secondary Outcome: Participant Systolic Blood Pressure Over Time
Description: Systolic blood pressure measures the pressure on the blood vessels when the heart is beats and thus is pushing blood to the rest of the body. A normal systolic blood pressure is lower than 120 mmHg. High blood pressure, as known as hypertension, is a risk factor for coronary artery disease, stroke, heart failure, and other complications if left unmanaged. The value closest to and within 6 weeks of the day expected was selected.
Time Frame: 26, 52, 104, 156, and 208 Weeks Post-Transplant
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
mmHg
  26 Weeks Post-Transplant | 131.5 [123 to 140]
  52 Weeks Post-Transplant: number analyzed (Participants) | 9
  52 Weeks Post-Transplant | 135 [130 to 140]
  104 Weeks Post-Transplant: number analyzed (Participants) | 6
  104 Weeks Post-Transplant | 137 [135 to 148]
  156 Weeks Post-Transplant: number analyzed (Participants) | 3
  156 Weeks Post-Transplant | 140 [120 to 140]
  208 Weeks Post-Transplant: number analyzed (Participants) | 4
  208 Weeks Post-Transplant | 132 [123.5 to 135]

20. Secondary Outcome: Participant Diastolic Blood Pressure Over Time
Description: Diastolic blood pressure measures the pressure in the arteries when the heart is at rest and is thus filled with blood. A normal diastolic blood pressure is lower than 80 mmHg. High blood pressure, as known as hypertension, is a risk factor for coronary artery disease, stroke, heart failure, and other complications if left unmanaged. The value closest to and within 6 weeks of the day expected was selected.
Time Frame: 26, 52, 104, 156, and 208 Weeks Post-Transplant
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
mmHg
  26 Weeks Post-Transplant | 77.5 [71 to 86]
  52 Weeks Post-Transplant: number analyzed (Participants) | 9
  52 Weeks Post-Transplant | 77 [74 to 88]
  104 Weeks Post-Transplant: number analyzed (Participants) | 6
  104 Weeks Post-Transplant | 79 [72 to 88]
  156 Weeks Post-Transplant: number analyzed (Participants) | 3
  156 Weeks Post-Transplant | 76 [58 to 92]
  208 Weeks Post-Transplant: number analyzed (Participants) | 4
  208 Weeks Post-Transplant | 73 [66.5 to 79.5]

21. Secondary Outcome: Participant Total Cholesterol Over Time
Description: Total cholesterol measures the amount of cholesterol found in the blood. Cholesterol is a waxy substance your body needs to build cells, but too much can be a problem since it can build-up in arteries. Narrowed arteries can result in heart attack or stroke. A value less than 200 mg/dL is considered good. The value closest to and within 12 weeks of the day expected was selected.
Time Frame: 26, 52, 104, 156, and 208 Weeks Post-Transplant
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
mg/dL
  26 Weeks Post-Transplant: number analyzed (Participants) | 8
  26 Weeks Post-Transplant | 188 [168 to 215.5]
  52 Weeks Post-Transplant: number analyzed (Participants) | 4
  52 Weeks Post-Transplant | 141.5 [129.5 to 170]
  104 Weeks Post-Transplant: number analyzed (Participants) | 8
  104 Weeks Post-Transplant | 165 [149 to 172]
  156 Weeks Post-Transplant: number analyzed (Participants) | 3
  156 Weeks Post-Transplant | 175 [153 to 199]
  208 Weeks Post-Transplant: number analyzed (Participants) | 3
  208 Weeks Post-Transplant | 173 [118 to 285]

22. Secondary Outcome: Participant Glucose Level Over Time
Description: This is a measure of glucose found in the blood. Glucose, a sugar, is an energy source that the body relies on to properly function. If levels are too high for a long period of time, diabetes can develop. Diabetes can result in many long-term complications such as eye, kidney, and nerve damage, stroke, and cardiovascular complications. Fasting levels for glucose should be around 70-99 mg/dL and less than 140 mg/dL within 2 hours after a meal. The value closest to and within 6 weeks of the day expected was selected.
Time Frame: 26, 52, 104, 156, and 208 Weeks Post-Transplant
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Induction (Rituximab and ATG)
Number analyzed (Participants) | 10
mg/dL
  26 Weeks Post-Transplant | 103.5 [96 to 112]
  52 Weeks Post-Transplant: number analyzed (Participants) | 9
  52 Weeks Post-Transplant | 108 [90 to 116]
  104 Weeks Post-Transplant: number analyzed (Participants) | 6
  104 Weeks Post-Transplant | 96.5 [83 to 129]
  156 Weeks Post-Transplant: number analyzed (Participants) | 4
  156 Weeks Post-Transplant | 104.5 [94 to 208]
  208 Weeks Post-Transplant: number analyzed (Participants) | 4
  208 Weeks Post-Transplant | 83.5 [75.5 to 141]

ADVERSE EVENTS:
Time Frame: Transplantation through end of trial participation (up to 4.4 years post-transplant).
Groups:
- Transplanted: These are adult living donor kidney transplant recipients that were enrolled into the study prior to transplant and met all criteria for study participation. These participants received a novel induction regimen of ATG and rituximab that included 4 doses of ATG 1.5 mg/kg and 2 doses of rituximab 375 mg/m2. The first dose of rituximab was given around day -6 prior to transplant, and the second dose was given on day 1-3 post-transplant. The first dose of ATG was given on the day of transplant, with the additional three doses administered on days 2-7 post-transplant (not on the same day as rituximab). Participants were maintained on the anti-rejection medications tacrolimus, MMF, and sirolimus after transplant. Participants were evaluated for eligibility to start gradual withdrawal of their anti-rejection medications starting as early as 26 weeks post-transplant. Eligible participants were gradually withdrawn from anti-rejection medication over a period of 68-104 weeks.
Arm/Group | Transplanted
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplanted (N=10)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Transplant rejection (Immune system disorders) | 4 (4)
Pyelonephritis (Infections and infestations) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplanted (N=10)
Leukopenia (Blood and lymphatic system disorders) | 2 (6)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Transplant rejection (Immune system disorders) | 2 (2)
BK virus infection (Infections and infestations) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1)
Viraemia (Infections and infestations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (4)
Eosinophil count increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (5)
Transaminases increased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
IgA nephropathy (Renal and urinary disorders) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Varicose vein (Vascular disorders) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The stopping rule for the incidence of rejection was met in December 2015, and enrollment was stopped in January 2016. After another rejection in May 2016, all participants were removed from protocol therapy and into reduced safety follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No